CLINICAL TRIAL: NCT00594100
Title: The Embolic Protection With Reverse Flow Study of the GORE Neuro Protection System in Carotid Stenting of Subjects At High Risk for Carotid Endarterectomy
Brief Title: GORE Embolic Protection With Reverse Flow
Acronym: EMPiRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPS 05-05
Record Dates: First submitted 2007-12-20; First posted 2008-01-15 (Estimated); Results first posted 2009-05-05 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery stenosis; embolic protection device; GORE Neuro Protection System; GORE Flow Reversal System; reverse flow; proximal occlusion device; GNPS; Parodi; EMPiRE; distal embolization; minimizing risks of CAS; PAES
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GFRS Pivotal Subjects (Experimental): All non-training subjects using the GORE Flow Reversal System for embolic protection during carotid artery stenting (all subjects other than first two subjects accounted for in Training Cases).
  Interventions: Device: GORE Flow Reversal System (GFRS)

INTERVENTIONS:
Device: GORE Flow Reversal System (GFRS) — Carotid artery angioplasty and stenting with embolic protection
  Other Names: Gore Neuro Protection System

SUMMARY:
To compare the 30-day safety and efficacy of the GORE Flow Reversal System when used with approved carotid stents to an Objective Performance Criterion derived from distal embolic protection studies.

DETAILED DESCRIPTION:
The GORE Flow Reversal System, manufactured by W. L. Gore & Associates, Inc., was developed as a proximal occlusion device to reverse the flow of blood in the carotid artery. It is designed to achieve embolic protection prior to crossing the lesion in the majority of cases in order to minimize the possibility of an adverse event occurrence.

The objective of this study is to assess the safety and effectiveness of the GORE Flow Reversal System when used to provide embolic protection during Carotid Artery Stent (CAS) procedures. Subjects diagnosed with carotid stenosis requiring revascularization and are at high risk for adverse events from CEA are eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Carotid stenosis requiring revascularization and indicating either symptomatic status, with carotid stenosis ≥ 50% OR asymptomatic status with carotid stenosis ≥ 80%
* Target lesion is located in one of the following:(a) internal carotid artery (ICA) (b) bifurcation (c) common carotid artery (CCA) proximal to the bifurcation
* At Anatomic risk for adverse events from CEA (e.g. restenosis after a prior CEA) OR at Co-morbid risk for adverse events from CEA (e.g., unstable angina with ECG changes)

Exclusion Criteria:

* Recent surgical procedure within 30 days before or after the stent procedure
* Uncontrolled sensitivity to contrast media
* Renal Insufficiency
* Recent evolving, acute stroke within 21 days of study evaluation
* Myocardial infarction within 72 hours prior to stent procedure
* History of a prior major ipsilateral stroke with residual neurological deficits likely to confound the neurological assessments (e.g., NIHSS)
* Neurological deficits not due to stroke likely to confound the neurological assessments (e.g., NIHSS)

Angiographic Exclusion Criteria:

* Isolated ipsilateral hemisphere leading to subject intolerance to reverse flow
* Total occlusion of the ipsilateral carotid artery
* Pre-existing stent in the ipsilateral carotid artery OR the contralateral carotid artery that extends into the aortic arch
* Presence of a filling defect, thrombus, occlusion or "string sign" in the target vessel
* Severe lesion calcification restricting stent deployment
* Carotid stenosis located distal to target stenosis that is more severe than target stenosis
* > 50% stenosis of the CCA proximal to target vessel
* Known mobile plaque in the aortic arch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clair, M.D., Principal Investigator — The Cleveland Clinic; L. N. Hopkins, M.D., Principal Investigator — Millard Fillmore Gates/Univ. of Buffalo
Locations (2):
- United States (2):
  - Millard Fillmore Gates/Univ. of Buffalo, Buffalo, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Background] Parodi JC. Re: is flow reversal the best method of protection during carotid stenting? J Endovasc Ther. 2005 Jun;12(3):414-5. doi: 10.1583/05-1610L.1. No abstract available. PMID 15943521
- [Background] Parodi JC, Schonholz C, Parodi FE, Sicard G, Ferreira LM. Initial 200 cases of carotid artery stenting using a reversal-of-flow cerebral protection device. J Cardiovasc Surg (Torino). 2007 Apr;48(2):117-24. PMID 17410059
- [Background] Parodi JC, Schonholz C, Ferreira LM, Mendaro E, Ohki T. "Seat belt and air bag" technique for cerebral protection during carotid stenting. J Endovasc Ther. 2002 Feb;9(1):20-4. doi: 10.1177/152660280200900104. PMID 11958320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was approved to enroll subjects from a maximum of 40 medical institutions in the United States (including public and academic research center hospitals and private practices).
Period: Procedure
Arm/Group | GFRS Pivotal Subjects
Started | 245
Completed | 236
Not Completed | 9
Not completed — Technical Failure | 9
Period: Follow-up Through 30 Days Post Procedure
Arm/Group | GFRS Pivotal Subjects
Started | 236
Completed | 224
Not Completed | 12
Not completed — Death / Reintervention / Medical Reasons | 2
Not completed — Discontinued Prior to Visit | 6
Not completed — Missed Visit - Phone Contact Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | GFRS Pivotal Subjects
Number analyzed (Participants) | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (9.6)
Age, Continuous [Median (Full Range); unit: years] | 71.0 [46.0 to 89.8]
Age, Customized [Number; unit: participants]
  < 80 years | 207
  >= 80 years | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 165
History of Diabetes [Number; unit: participants] — Patient has a history of Diabetes prior to enrollment
  participants
    Yes | 86
    No | 159
History of Hypertension [Number; unit: participants] — Patient has history of hypertension prior to study enrollment
  participants
    Yes | 212
    No | 33
History of Ischemic Stroke [Number; unit: participants] — Number of prior ischemic strokes prior to enrollment
  participants
    None | 192
    One | 42
    Two or More | 11
Previous Endarterectomy [Number; unit: participants] — Timing of previous endarterectomy (CEA)
  participants
    None | 143
    Less than 1 Year | 23
    Greater than 1 Year | 79
Symptomatic [Number; unit: participants] — Presence of baseline neurological symptoms within 6 months prior to study enrollment
  participants
    Symptomatic | 78
    Asymptomatic | 167

OUTCOME MEASURES:

1. Primary Outcome: Composite Major Adverse Event (MAE) Rate
Description: Number of participants with one or more Major Adverse Event (death, stroke, myocardial infarction, and/or transient ischemic attack (TIA)) through the 30-day follow-up (non-hierarchical; MAE adjudicated by independent Clinical Events Committee)
Time Frame: Treatment through 30-day visit window
Population: All primary endpoint evaluable subjects
Measure: Number; unit: participants
Arm/Group | GFRS Pivotal Subjects
Number analyzed (Participants) | 202
participants
  Major Ischemic Stroke | 0
  Minor Ischemic Stroke | 5
  Hemorrhagic Stroke | 2
  Death | 2
  Death / Any Stroke | 7
  Myocardial Infarction (MI) | 2
  Death / Stroke / MI | 9
  Transient Ischemic Attack (TIA) | 2
  Overall MAE | 11
Statistical Analysis 1: Comparison: GFRS Pivotal Subjects; The EMPiRE Study tested the null hypothesis that the true MAE rate was greater than or equal to an Objective Performance Criterion (OPC) of 11.83% versus the alternative hypothesis that the true MAE rate was less than the OPC. The sample size was calculated based on 80% power and a Type I error rate of 0.025. The OPC was calculated from results of published carotid artery stenting studies that utilized distal embolic protection systems; Test type: Superiority or Other; p = 0.002, One-Sample Binomial; Significance test was based on a one-sample binomial test; Binomial Proportion = 0.054, 95% CI 2-sided [0.027 to 0.095], Standard Error of Mean 0.016 — 95% Confidence Interval is exact binomial using Clopper-Pearson method. Standard Error is from Normal approximation

2. Secondary Outcome: Flow Reversal System Technical Success
Description: Number of participants with Technical Success using the GORE Flow Reversal System (system deployed and utilized during stenting procedure)
Time Frame: Procedure
Population: All enrolled subjects
Measure: Number; unit: participants
Arm/Group | GFRS Pivotal Subjects
Number analyzed (Participants) | 245
participants | 236

3. Secondary Outcome: Flow Reversal System Success
Description: Number of participants where the GORE Flow Reversal System was delivered, placed, reverse flow was established, and the balloon sheath and wire retrieved as outlined in the Instructions for Use without causing any adverse events during the procedure.
Time Frame: Procedure
Measure: Number; unit: participants
Arm/Group | GFRS Pivotal Subjects
Number analyzed (Participants) | 245
participants | 233

4. Secondary Outcome: Stent Success
Description: Number of participants where the FDA-approved stent was successfully delivered, deployed,and delivery system removed with an attainment of < 50% residual stenosis following stent placement, as assessed by the angiographic core laboratory.
Time Frame: Procedure
Population: All enrolled subjects with post procedure angiographic assessment of lesion stenosis
Measure: Number; unit: participants
Arm/Group | GFRS Pivotal Subjects
Number analyzed (Participants) | 230
participants | 228

5. Secondary Outcome: Clinical Success
Description: Number of participants with Flow Reversal System and Stent Success in the absence of death, emergency endarterectomy, repeat percutaneous transluminal angioplasty (PTA)/thrombolysis of the target vessel, stroke, or myocardial infarction (MI), as determined by the Clinical Events Committee (CEC).
Time Frame: 24-48 Hours Post-Procedure
Population: All enrolled subjects with post procedure angiographic assessment of lesion stenosis
Measure: Number; unit: participants
Arm/Group | GFRS Pivotal Subjects
Number analyzed (Participants) | 230
participants | 211

6. Secondary Outcome: Patency at 30 Days
Description: Number of participants with less than 50% restenosis as determined by carotid duplex ultrasound core laboratory at 30 days post-procedure.
Time Frame: Treatment through 30-day visit window
Population: Subjects with successful stent placement and ultrasound evaluation at 30-day follow-up evaluation.
Measure: Number; unit: participants
Arm/Group | GFRS Pivotal Subjects
Number analyzed (Participants) | 186
participants | 182

ADVERSE EVENTS:
Time Frame: 30 days postprocedure (0-40 days given 10-day late follow-up window)
Description: AEs reported by investigative sites via Adverse Event Case Report Form (CRF), using study-specific coding. Site-reported adverse events that were potential Major Adverse Events (stroke or TIA) were adjudicated by the independent Clinical Events Committee.
Arm/Group | GFRS Pivotal Subjects
Serious Adverse Events (participants affected / at risk) | 40/245
Other Adverse Events (participants affected / at risk) | 62/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFRS Pivotal Subjects (N=245)
Hypotension (Cardiac disorders) | 14 (14)
Groin Hematoma (w/wo Surgical Repair) (Blood and lymphatic system disorders) | 2 (2)
Other (Bleeding) (Blood and lymphatic system disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Angina/Coronary Ischemia (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 4 (4)
Congestive Heart Failure (CHF) (Cardiac disorders) | 1 (1)
Myocardial Infarction (MI) (Cardiac disorders) | 3 (3)
Stroke/Cerebrovascular accident (CVA) (Nervous system disorders) | 5 (5)
Cerebral ischemia/Transient ischemic attack (TIA) (Nervous system disorders) | 1 (3)
Other (Cardiac) (Cardiac disorders) | 4 (4)
Renal Failure/Insufficiency (Renal and urinary disorders) | 1 (1)
Other (Infectious/Inflammatory) (Infections and infestations) | 3 (3)
Other (Neurologic) (Nervous system disorders) | 2 (3)
Hyperperfusion Syndrome (Nervous system disorders) | 1 (1)
Pain (Head, Neck) (Nervous system disorders) | 1 (1)
Other (Surgical Procedure) (Surgical and medical procedures) | 1 (1)
Pseudoaneurysm (Femoral) (Vascular disorders) | 1 (1)
Other (Wound) (Injury, poisoning and procedural complications) | 1 (1)
Other (Other) (General disorders) | 5 (6)
Cerebral Hemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFRS Pivotal Subjects (N=245)
Arrhythmia (Cardiac disorders) | 8 (8)
Hypotension (Cardiac disorders) | 28 (28)
Hypertension (Cardiac disorders) | 12 (13)
Other (Neurologic) (Nervous system disorders) | 9 (11)
Pain (Head, Neck) (Nervous system disorders) | 11 (11)
Other (Other) (Surgical and medical procedures) | 18 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.